CLINICAL TRIAL: NCT00190593
Title: Raloxifene Hydrochloride or Placebo in Postmenopausal Women at Risk for Major Coronary Events
Brief Title: Raloxifene Use for The Heart
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1865; H3S-MC-GGIO
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Cardiovascular Diseases; Breast Neoplasms
MeSH Terms: conditions — Cardiovascular Diseases; Breast Neoplasms | interventions — Raloxifene Hydrochloride

INTERVENTIONS:
Drug: raloxifene
Drug: placebo

SUMMARY:
The purpose of this study is to determine whether raloxifene compared with placebo lowers the risk of coronary events and reduces the risk of invasive breast cancer in postmenopausal women at risk for major coronary events.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with established coronary heart disease or at risk for a major coronary event.

Exclusion Criteria:

* Postmenopausal symptoms that required estrogen replacement therapy.
* Suspected or known history of breast or endometrial carcinoma.
* Known or probable history of deep venous thrombosis, pulmonary embolism, or retinal vein thrombosis.
* New York Heart Association classes III or IV heart failure.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000
Dates: Start 1998-06; Study Completion 2005-11

PRIMARY OUTCOMES:
Time to first occurrence of coronary death, non-fatal myocardial infarction (MI), or hospitalized acute coronary syndrome other than MI combined after an expected 5 to 7.5 years of follow-up.
Time to first occurrence of invasive breast cancer after an expected 5 to 7.5 years of follow-up.

SECONDARY OUTCOMES:
After an expected 5 to 7.5 years of follow-up:
Cardiovascular death, non-fatal MI, hospitalized acute coronary syndrome other than MI, myocardial revascularization, and stroke (individually and combined)
All-cause hospitalization and mortality
Non-coronary artery revascularization
Non-traumatic lower extremity amputation
Fractures
Venous thromboembolism.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additonal information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Wenger NK, Barrett-Connor E, Collins P, Grady D, Kornitzer M, Mosca L, Sashegyi A, Baygani SK, Anderson PW, Moscarelli E. Baseline characteristics of participants in the Raloxifene Use for The Heart (RUTH) trial. Am J Cardiol. 2002 Dec 1;90(11):1204-10. doi: 10.1016/s0002-9149(02)02835-7. PMID 12450599
- [Background] Mosca L, Barrett-Connor E, Wenger NK, Collins P, Grady D, Kornitzer M, Moscarelli E, Paul S, Wright TJ, Helterbrand JD, Anderson PW. Design and methods of the Raloxifene Use for The Heart (RUTH) study. Am J Cardiol. 2001 Aug 15;88(4):392-5. doi: 10.1016/s0002-9149(01)01685-x. PMID 11545760
- [Result] Barrett-Connor E, Mosca L, Collins P, Geiger MJ, Grady D, Kornitzer M, McNabb MA, Wenger NK; Raloxifene Use for The Heart (RUTH) Trial Investigators. Effects of raloxifene on cardiovascular events and breast cancer in postmenopausal women. N Engl J Med. 2006 Jul 13;355(2):125-37. doi: 10.1056/NEJMoa062462. PMID 16837676
- [Derived] Daniels LB, Grady D, Mosca L, Collins P, Mitlak BH, Amewou-Atisso MG, Wenger NK, Barrett-Connor E; Raloxifene Use for the Heart (RUTH) Trial Investigators. Is diabetes mellitus a heart disease equivalent in women? Results from an international study of postmenopausal women in the Raloxifene Use for the Heart (RUTH) Trial. Circ Cardiovasc Qual Outcomes. 2013 Mar 1;6(2):164-70. doi: 10.1161/CIRCOUTCOMES.112.966986. Epub 2013 Mar 12. PMID 23481531
- [Derived] Collins P, Mosca L, Geiger MJ, Grady D, Kornitzer M, Amewou-Atisso MG, Effron MB, Dowsett SA, Barrett-Connor E, Wenger NK. Effects of the selective estrogen receptor modulator raloxifene on coronary outcomes in the Raloxifene Use for The Heart trial: results of subgroup analyses by age and other factors. Circulation. 2009 Feb 24;119(7):922-30. doi: 10.1161/CIRCULATIONAHA.108.817577. Epub 2009 Feb 9. PMID 19204301